CLINICAL TRIAL: NCT02777892
Title: Pulmonic SAPIEN S3™ THV Registry A Multi-center, Observational Registry With Retrospective Enrollment of Patients That Underwent Transcatheter Pulmonic Valve Implantation and a Retrospective or Prospective Follow-up
Brief Title: Pulmonic SAPIEN S3™ THV Registry
Acronym: PulmonicS3
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: Pulmonic S3
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Valve Malfunction; Right Ventricular Outflow Tract (RVOT) Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary valve replacement: SAPIEN S3 Transcatheter Heart Valve in the pulmonic position at the time of data collection
  Interventions: Other: Sapien S3

INTERVENTIONS:
Other: Sapien S3 — Patients that have undergone percutaneous implantation of an Edwards SAPIEN S3 Transcatheter Heart Valve in the pulmonic position at the time of data collection

SUMMARY:
Multi-center, Observational Registry with Retrospective Enrollment and Prospective Follow-up.

The aim of the registry is to document the feasibility and safety of implanting an Edwards SAPIEN S3 transcatheter heart valve in the pulmonic position

DETAILED DESCRIPTION:
A malfunction or dysplasia of the pulmonary valve or the right ventricular outflow tract (RVOT) is one of the major components of the cardiac physiology in many congenital heart defects. Surgical correction of complex heart defects often includes some form of surgical repair or replacement of the native RVOT by biological valves such as homograft, bioprosthesis or Xenografts (i.e., Contegra conduits). Typical examples are tetralogy of Fallot (TOF) or double outlet right ventricle (DORV), pulmonary stenosis (PS), pulmonary atresia (PA), truncus arteriosus (TA), transposition of the great arteries (TGA) with PS (Rastelli's operation), absent pulmonary valve syndrome (Miller-Lev-Paul), Ross surgery for aortic valve disease and others. The repaired or replaced pulmonary valve however often becomes dysfunctional later on and many patients require surgical revisions of the RVOT with pulmonary valve replacement within 10 years of primary intervention.

TPVI provides a less invasive alternative to surgery in patients with right ventricular-to-pulmonary artery (RV-PA) conduit dysfunction. Early results of percutaneous pulmonary valve implantation (PPVI) showed that it is a promising procedure compared to a conventional surgical intervention. Meanwhile, pre-stenting of the RVOT before PPVI is routinely performed, enabling PPVI in various anatomies.

ELIGIBILITY:
Inclusion criteria

* Clinical indication and decision for the implantation of an Edwards SAPIEN 3 THV made
* Data release form

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have undergone percutaneous implantation of an Edwards SAPIEN XT Transcatheter Heart Valve in the pulmonic position at the time of data collection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
changes in right ventricular and pulmonary artery pressure | from baseline to 30 days after implantation

SECONDARY OUTCOMES:
Max. flow velocity RVOT | 30 days after implantation
Changes in NYHA class | from baseline to 30 days after implantation
changes in degree of pulmonary regurgitation | from baseline to 30 days after implantation
length of hospitalization | 30 days after implantation
changes in Peak Oxygen consumption | from baseline to 24 months after implantation
Percentage of cases with proper device function | 24 months after implantation
Incidence of structural valve Deterioration including stent fracture | 24 months after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bramlage, Prof MD, Study Director — Institut für Pharmakologie und Präventive Medizin
Locations (4):
- St Pauls Hospital Vancouver, Vancouver, British Columbia, Canada
- Germany (2):
  - Deutsches Herzzentrum München, München, Bavaria
  - Herzchirurgische Klinik und Poliklinik LMU, München, Bavaria
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: on-line data entry site — https://ippmed-pulmonics3.s4trials-europe.net